CLINICAL TRIAL: NCT02309034
Title: Aquatic and Land Physical Training Effects on Cardiometabolic Risk Factors in Adolescents With Overweight and Obesity: a Randomized Controlled Clinical Trial.
Brief Title: Aquatic and Land Physical Training Effects on Cardiometabolic Risk Factors in Adolescents With Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 140485
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Cardiometabolic risk factors; Adolescents; Exercise
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Aquatic Therapy; Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Jump exercise (Experimental): rebound exercises.
  Interventions: Behavioral: Jump exercise; Other: Nutritional guidance
- Aquatic exercise (Experimental): Hydrogimnastic.
  Interventions: Behavioral: Aquatic exercise; Other: Nutritional guidance
- Nutritional guidance (Active Comparator): Nutritional counseling classes.
  Interventions: Other: Nutritional guidance

INTERVENTIONS:
Behavioral: Jump exercise — Land Group / Jump (LG): Will hold weekly classes of nutritional guidance and three weekly sessions of jump, for 12 weeks, divided into warm up, main aerobics and relaxation.
  Other Names: Rebound exercises
  Arms: Jump exercise
Behavioral: Aquatic exercise — Group Water / Water aerobics (WG): Will hold weekly classes of nutritional guidance and three weekly sessions of water, for 12 weeks, divided into warm up, main aerobics and relaxation.
  Other Names: Hydrogimnastic
  Arms: Aquatic exercise
Other: Nutritional guidance — Control Group (CG): take part only of weekly classes of nutritional guidance, in addition to a closed group on Facebook in order to encourage them and increase attention to the group.
  Other Names: Nutritional counseling

SUMMARY:
Objective: To compare the results of two types of low-impact exercise training, in and out of the water, with the control group, regarding cardiometabolic risk factors in overweight adolescents; and to investigate the changes resulting from interventions in biochemical, anthropometric, psychological variables and body composition.

Experimental design: Randomized clinical trial with overweight and obesity adolescents.

Local Search: College of Physical Education of Federal University of Rio Grande do Sul and Hospital de Clinicas de Porto Alegre, city of Porto Alegre, Rio Grande do Sul State, Brazil.

Participants: Took part in the study 75 overweight and obesity adolescents, pubertal and post-pubertal, recruted by announcement in the most important newspapers of Porto Alegre city.

Intervention: Adolescents that acepted to participate in the study, and authorized by their parents, were randomized into three groups: Group Land / Jump, with three weekly sessions Jump; Water / hidrogimnastic group, with three weekly sessions of hidrogminastic; Control group that not participate in physical exercise intervention. The intervention will last 12 weeks and three groups participate in weekly sessions of nutritional guidance. Assessments occur at the beginning of the intervention program and 72 hours after the 12th week of the program. The results of all study variables among the three groups in the two time points, and in each group between the two periods, will compared.

Measures: Anthropometric, biochemical and blood pressure evaluations, in addition to applying instruments for assessing quality of life, body image and mental health by experienced evaluators, as well as blood draws conducted by an experienced gatherer's Hospital de Clínicas de Porto Alegre.

Expected Results: In the study, are been expected to verify that the exercise programs, aquatic and land, associated with nutritional guidance, are efficient to modify positively the outcomes studied.

DETAILED DESCRIPTION:
Methods:

The sample will be selected intentionally with 75 subjects. Those who agree to participate in the study will be randomly allocated into three groups by a blinded evaluator for the study, which will use online www.randomizer.org the software as follows: aqua + nutritional counseling, jump + nutritional counseling, group control (nutritional counseling only), all with 12-week duration.

The study examine the effects obtained by the three groups on outcomes of cardiometabolic risk factors (waist circumference, blood pressure, HDL-cholesterol, triglycerides, fasting glucose), outcomes of amount and distribution of body fat (sum of skinfolds - triceps subscapular, suprailiac, abdominal and mid thigh - by bioelectrical impedance body fat percentage and waist / height), and psychological variables (quality of life, body image and mental health). In addition, nutritional counseling at weekly sessions will be used as a control variable. Characterization data of the sample (age, sex, weight, height, and waist / height) and other biochemical endpoints also comprise the study (total cholesterol, LDL-cholesterol, fasting insulin, HOMA-IR, QUICK, and high-sensitivity C- reactive protein will be collected).

All measurements follow standard and validated procedures for the population object of study.

To the chronic effect analysis, blood samples will be collected two times, before and after training period, with 12 hours fasting. To avoid the acute effect of the exercises, the measurements will done 72 hours after the 12th week.

A sample of 5 ml of blood per antecubital vein will collected. The sample will be collected at the school for experienced gatherer, and will be taken immediately to the laboratory in order to ensure that analyzes are performed on the same day.

The health-related quality of life will assessed using the questionnaire on pediatric quality of life PedsQL 4.0, adolescents and their parents.

For analysis of body satisfaction instrument Body Shape Questionnaire BSQ will used. To ascertain the perception of body image will applied to Scale Silhouettes of Stunkard.

Mental health will assessed using the Strengths and Difficulties Questionnaires SDQ.

For classification of maturational stage, will held assessment of sexual maturation stages proposed by Tanner, determined by self-assessment of the stage of development of pubic hair, avoiding major constraint adolescents.

Intervention with exercise:

The groups will perform physical training activities three times a week after school for 12 weeks, with interval training sessions varying intensities according to the scale of perceived exertion Borg, with duration ranging between 24 and 32 minute main part. Classes will taught by a physical education teacher with the aid of monitors, area students.

Nutrition education classes will held at the school, by nutritionist, with a weekly, totaling 12 meetings.

Training Protocol Both trainings will be conducted simultaneously with each group in their midst, in order to avoid possible interference on the voice command, ambient temperature, relative humidity and time of accomplishment from training.

ELIGIBILITY:
Inclusion Criteria:

* Pubescent and post-pubescent adolescents are included, of both gender, who have overweight or obese, and waist / height ratio greater than 0.50
* Without disabling the practice of physical exercise conditions and not using medications that may affect the outcome of the present study, such as medications to control cholesterol for hormone treatments and diuretics

Exclusion Criteria:

* Those adolescents who become pregnant during the training will be deleted

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | baseline, 12th week

SECONDARY OUTCOMES:
Waist circumference | baseline, 12th week
Blood Pressure | baseline, 12th week
HDL-cholesterol | baseline, 12th week
Triglycerides | baseline, 12th week
Fasting glycemia | baseline, 12th week
Body Fat Percentage | baseline, 12th week
  Bioeletrical Impedance

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz D Schaan, PhD, Principal Investigator — Federal University of Rio Grande do Sul